CLINICAL TRIAL: NCT06018233
Title: The Role Of Technology In Addressing Societal Challenges: A New Regime For The Law And Governance Of Innovation
Brief Title: Role of Technology in Addressing Societal Challenges - New Governance
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-010-23
Record Dates: First submitted 2023-08-11; First posted 2023-08-30 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Power
Keywords: Governance; Technology; Data; Intersection; Intellectual Property; Regulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People involved with creating and operating regimes which address key societal challenges.: Qualitative semi-structured interviews to explore approaches taken to regimes, including one case study group regarding the Public Benefit and Privacy Panel in Scotland. No use of drugs and no personal health related interventions. Same approaches taken to 3 other case study groups which do not involve health.
  Interventions: Other: New proposal for regime creation

INTERVENTIONS:
Other: New proposal for regime creation — Interviews and building of proposals in the light of the information obtained and desk based research

SUMMARY:
Technology and data can bring opportunities for increased societal benefits for example regarding health, environmental sustainability and energy. There can be clashes between regimes which aim to bring these benefits about, and the outcomes which are dictated if one looks to only laws and regimes with a focus on technology and data, notably information and intellectual property (IP) laws. A recent example of a clash was seen between IP, human rights and health in relation to COVID-19.

This study is part of a project exploring the place and impact of clashes on the operation of regimes and possible new potential forms of governance, structure and regime creation which could be developed. The project will explore the establishment and operation of the Scottish Public Benefit and Privacy Panel for Health and Social Care. It will also explore approaches to data and technology in the UK oil and gas licensing framework; a developing new international regime in relation to marine biodiversity, benefit sharing and technology transfer; and approaches in Scotland and in England to private or public ownership and licensing of soil and environmental data, including those funded by research councils. It may also include the European data strategy and the development of the pan African free trade agreement and its approach to IP. Some of these regimes engage directly with laws relating to data and technology, notably private rights, information control and IP; some do not.

The study will interrogate, through qualitative research with key figures who and are involved, the drivers for structural approaches being taken; levels of engagement in creating and operating new regimes with regime and laws focussed on data and technology; and the possible impact of data and technology regimes on the new regimes' wider goals.

DETAILED DESCRIPTION:
The project explores the different frameworks, and the possible consequences of limited engagement with data and technology, for delivery of the ultimate societal goals. Proposals are then developed for more holistic and pluralist engagement when new regimes, in their different forms, are created.

This project will make an important contribution to scholarship regarding legal policy making, governance, regulation, legal theory, pluralism, private and public intersections and "wicked problems". The findings of this project will be of value to scholars, policy makers and activists in developing a more open and informed approach to choices which could be made, means by which they could be delivered, and to reaching more effective solutions to address societal challenges through a lens - direct or indirect - of data and technology.

The project's principal objective is to develop new theoretical approaches and practical paths which could be applied, at national and international level, substantively and structurally, to creating and operating regimes which address key societal challenges using data and technology.

The project's proposals will enable decision makers - irrespective of subject matter or starting point - to take a wide view of relevance, to engage widely with stakeholders and experts and to see nothing as unchallengeable or as the responsibility of another regime. The project will also explore the extent to which a hierarchy or overarching common goals could be created, such as stewardship and respect for the commons (or indeed private property), within which governance of data, technology and also ultimate societal goals could and should be delivered.

Much of the project is based on theory and desk based reviews of scholarship and of publicly available sources. It will consider legislation, treaties, case law, policy and activist work and governance and regulatory frameworks. It will engage with ongoing developments in judicial innovation, interpretation of legislation and application of regulatory approaches, notably regarding precaution and certainty. It will draw on the intersection between law, philosophy and science and the extent to which different approaches could and should be taken to rawer information and that which has been the subject of processing and refinement.

Complementing this, the study will carry out semi-structured qualitative interviews with research participants.

Interviews will be carried out online via TEAMS, and the interviews will be recorded using an encrypted dictaphone and then transcribed by the researcher. Before the transcribing is carried it, each participant will be accorded a legend (eg participant 1) and the transcript will be prepared on this basis. The transcripts will be provided to the interviewees via TEAMS in private subchannels for confirmation of accuracy before the data analysis stage commences.

Research participants will be individuals involved in creating and operating the regimes which are used as case studies. Abbe Brown anticipates interviewing each research participant once, although she will indicate that if future issues arise she may ask to speak to them again if they would be willing to do so, for clarification purposes.

Then, the data analysis phase will involve key word analysis of the transcripts based on questions asked, issues explored in the book, and from points arising in interview, in a grounded theory approach.

ELIGIBILITY:
Inclusion Criteria:

* involved in the development or operation of one of the relevant governance and regime structures listed.
* able to communicate in English
* no communication needs.
* able to give informed consent.

Exclusion Criteria:

* not involved in the development or operation of one of the relevant governance and regime structures listed.
* unable to communicate in English
* has communication needs
* is unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 - People involved in creation and operation of Scottish panel to grant access to data for re-use in health and social care research (Public Benefit and Privacy Panel for Health and Social Care of NHS Scotland).
  Group 2 - People involved in creation and operation of approaches to data and technology in a UK framework based on the grant of an oil and gas licence.
  Group 3 - People involved in developing new international regime in relation to marine biodiversity, benefit sharing and technology transfer.
  Group 4 - People involved in creation and operation of different approaches in Scotland and in England to private or public ownership and licensing of soil and environmental data, including those funded by a research council.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
New approaches to regime creation | 2 years 6 months project as whole. Interview phase as a whole, 4 months, each interview 1 hour, possible follow up.
  Interviews carried out, transcribed and shared with individual participants. Thereafter, by researcher, analysed, and considered although theoretical research. Proposals developed for more holistic and pluralist engagement and book written

CONTACTS AND LOCATIONS:
Overall Officials: Miss King, Study Director — University of Aberdeen and NHS Grampian
Locations (1):
- University of Aberdeen, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No